CLINICAL TRIAL: NCT03860428
Title: Randomized Non-inferiority Trial of Early Treatment Versus Expectant Management of Patent Ductus Arteriosus in Preterm Infants
Brief Title: Early Treatment Versus Expectant Management of PDA in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lviv National Medical University (Other)
Responsible Party: Principal Investigator, Dmytro Dobryanskyy, Clinical Professor, Lviv National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04011994
Record Dates: First submitted 2019-02-16; First posted 2019-03-04 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; Ibuprofen; Paracetamol; Expectant management
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen; Cyclooxygenase Inhibitors; Acetaminophen; Watchful Waiting; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rectal ibuprofen (Active Comparator): Early treatment of PDA that starts within the first 3 days of life using rectal ibuprofen q24h for 3 days, dosages: 20 mg/kg + 10 mg/kg + 10 mg/kg
  Interventions: Drug: Ibuprofen
- Intravenous paracetamol (Active Comparator): Early treatment of PDA that starts within the first 3 days of life using intravenous paraceta-mol 15 mg/kg q6h for 3 days
  Interventions: Drug: Paracetamol
- Expectant Treatment (Sham Comparator): Expectant PDA management is characterized as 'watchful waiting'. No intervention is initiated with the intention to close a PDA unless defi-nitely needed based of the predefined infant's condition.
  Interventions: Other: Expectant Management

INTERVENTIONS:
Drug: Ibuprofen — In the medical treatment arm the in-tention is to close the ductus arteriosus.
  Other Names: Cyclooxygenase Inhibitor
  Arms: Rectal ibuprofen
Drug: Paracetamol — In the medical treatment arm the in-tention is to close the ductus arteriosus.
  Other Names: Infulgan, Acetaminophen
  Arms: Intravenous paracetamol
Other: Expectant Management — Expectative PDA management is character-ized as 'watchful waiting'. No intervention is initiated with the intention to close a PDA.
  Other Names: Conservative management
  Arms: Expectant Treatment

SUMMARY:
Patent ductus arteriosus (PDA) in very preterm newborns is associated with severe neonatal mor-bidity: intraventricular hemorrhage (IVH), bronchopulmonary dysplasia (BPD), necrotizing en-terocolitis (NEC), retinopathy of prematurity (ROP). Existing methods of management PDA do not reduce the incidence of these diseases. The efficacy of cyclooxygenase inhibitors (COX) which are currently the standard of treatment in extreme preterm infants is about 70-80%. COX inhibitors have significant side effects. On the other hand, surgical ligation of the ductus arteriosus is associated with deterioration due to cardio-pulmonary problems and long-term complications. Paracetamol has been proposed for treatment of hemodynamically significant PDA because it has a different mecha-nism of action compared with COX inhibitors and a better safety profile.

Recently, expectant approach has becoming more popular, although there is not enough evidence to support it.

The objective of this study is to investigate whether in preterm infants, born at a GA less than 32 weeks, with a PDA (diameter > 1.5 mm) at a postnatal age of < 72 h, an expectant management is non-inferior to early treatment with regard to the composite of mortality and/or severe morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 weeks
* Birthweight <1500 g
* Age less than 72 hours
* PDA diameter > 1.5 mm
* Signed informed consent obtained from both parents

Exclusion Criteria:

* Birthweight ≥ 1500 g and/or gestation age ≥ 32 weeks
* Lack of informed consent of the parents
* Congenital heart defect, other than PDA and/or patent foramen ovale (PFO)
* The presence of a clinically apparent hemorrhagic syndrome
* Any intraventricular hemorrhage (IVH) in the first 48 hours or IVH grade 3-4
* A platelet count of < 50,000/mm3
* A serum creatinine concentration of > 110 μmol/L
* Oliguria <1 ml/kg/h
* Suspected/apparent NEC
* Suspected/apparent lung hypoplasia

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of bronchopulmonary dysplasia (BPD) or mortality at 36 weeks postmenstrual age (PMA) | 36 weeks PMA

SECONDARY OUTCOMES:
PDA re-opening rate | Day 1 up to 3 month
  PDA re-opening after echocardiographically documented closure
Closure rate of PDA within a week after the first and second course of pharmacological treatment | Participants will be evaluated at the end of first and second course, at an expected avarage of 10 days of life
The need for surgical ductus closure | Day 1 up to 3 month
Duration of any ventilation assist | Day 1 up to 3 month
  The ventilation assist time period
Duration of oxygen supplementation | Day 1 up to 3 month
  Days on supplement oxygen
Age of administration of full volume of enteral nutrition | Day 1 up to 3 month
Incidence of oliguria | In the first 14 days of life
Incidence of hypotension | Day 1 up to 3 month
Incidence of BPD | 36 weeks PMA
Mortality rate | 36 weeks PMA
Incidence of severe intraventricular hemorrhage | 28-days since birth
Incidence of necrotizing enterocolitis (Bell stage ≥ IIa) | 36 weeks PMA
Incidence of periventricular leukomalacia | 36 weeks PMA

CONTACTS AND LOCATIONS:
Overall Officials: Dmytro Dobryanskyy, MD, PhD, Principal Investigator — L'viv National Medical University
Locations (1):
- Lviv National Medical University, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Potsiurko S, Dobryanskyy D, Sekretar L. Patent ductus arteriosus, systemic NT-proBNP concentrations and development of bronchopulmonary dysplasia in very preterm infants: retrospective data analysis from a randomized controlled trial. BMC Pediatr. 2021 Jun 19;21(1):286. doi: 10.1186/s12887-021-02750-9. PMID 34147090